CLINICAL TRIAL: NCT05242640
Title: Understanding Components of Mind-body Exercise for Physical Activity Engagement in Metabolic Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Kristen Kraemer, Instructor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 2022P000037
Record Dates: First submitted 2022-01-27; First posted 2022-02-16 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Mindful attention (Experimental): 16 sessions over 8 weeks (2x/week) of mindful attention audio recordings delivered via headphones
  Interventions: Other: Mindful attention
- Exercise (Experimental): 16 sessions over 8 weeks (2x/week) of moderate-intensity treadmill walking
  Interventions: Other: Exercise
- Exercise with mindful attention (Experimental): 16 sessions over 8 weeks (2x/week) of moderate-intensity treadmill walking utilizing mindful attention audio recordings delivered via headphones
  Interventions: Other: Exercise with mindful attention
- No intervention (No Intervention): No intervention sessions

INTERVENTIONS:
Other: Mindful attention — Participants will listen to mindful attention audio recordings via headphones
  Arms: Mindful attention
Other: Exercise — Participants will complete a moderate-intensity walking program
  Arms: Exercise
Other: Exercise with mindful attention — Participants will complete a moderate-intensity walking program while listening to mindful attention audio recordings via headphones
  Arms: Exercise with mindful attention

SUMMARY:
The aim of this study is to assess the feasibility and acceptability (e.g., enrollment, adherence, retention, acceptability of procedures and interventions) of a pilot factorial study design that will help elucidate components of mind-body exercise interventions. The study involves completing a walking program, a mindful attention program, a walking program that includes mindful attention, or no program at all. A "pilot" study is a smaller study that helps researchers to understand whether the study design can be carried out and what participants think about the study.

ELIGIBILITY:
Inclusion Criteria:

* Metabolic syndrome, defined as meeting 3 or more of the following criteria in the last 12 months at the time of medical record review: (a) BMI ≥ 25; (b) fasting glucose ≥ 100 [5.6 mmol/L] or A1C ≥ 5.7 or medications; (c) blood pressure ≥ 130 systolic or ≥ 85 diastolic or medications; (d) triglycerides ≥ 150 or 1.7 mmol/L or medications; (e) or HDL < 40mg/ dL for men and 50mg/dL for women or medications;
* insufficiently active, defined as a score ≤ 23 (moderate-to-strenuous units) on Godin-Shepard Leisure-Time Physical Activity Questionnaire;
* age 18-70 years;
* given medical clearance for moderate-intensity exercise and exercise stress testing by their primary care physician (PCP);
* access to a device with internet and videoconferencing capabilities

Exclusion Criteria:

* current diagnosis of any of the following: (a) coronary artery disease or other chronic heart diseases (e.g., heart failure) in which exercise would be contraindicated or that would preclude HRV analyses (e.g., some arrhythmias); (b) any diabetes; (c) chronic obstructive pulmonary disease or other severe lung dysfunction (e.g., severe asthma); (d) severe cognitive impairment
* >2 self-reported classes or self-guided mindfulness or mindful movement sessions per week in past 3 months
* self-reported inability to speak and read in English
* current beta blocker or calcium channel blocker medication
* uncontrolled hypertension, defined as resting blood pressure ≥ 150 systolic or ≥ 90 diastolic in the last 6 months
* self- or physician-reported contraindications for exercise (e.g., severe balance impairment, musculoskeletal restrictions)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2025-11-28 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of screening: screened to eligible ratio | Through study completion, an average of 1 year
  percent of screened individuals that were determined eligible for the study
Feasibility of enrollment: eligible to enrollment ratio | Through study completion, an average of 1 year
  percent of eligible individuals that enroll in the study; determined to be feasible if greater than or equal to 70% of eligible patients enroll
Feasibility of retention: retention at each assessment | 6 months
  percent of enrolled participants retained at post-intervention and 3-month follow-up; determined to be feasible if greater than or equal to 70% retention at each assessment
Feasibility of interventions: attendance rates for each session | 6 months
  percent session attendance; determined to be feasible if participants attend greater than or equal to 75% of sessions
Feasibility of survey completion: survey completion rates at each assessment | 6 months
  percent of participants that complete surveys at post-intervention and 3-month follow-up
Acceptability of interventions | 6 months
  Acceptability of the interventions will be assessed via overall satisfaction (1 = not at all to 10 = very much); determined to be acceptable if mean rating is greater than or equal to 7.5 across 80% of sessions
Acceptability of study design | 6 months
  Acceptability of the study design will be assessed via acceptability of study procedures (1= not at all to 10 = very much); determined to be acceptable if mean rating is greater than or equal to 7.5 across 80% of sessions
Perspectives on study interventions | Post-intervention (after 8 week intervention)
  Perspectives on study interventions will be assessed via exit interview

SECONDARY OUTCOMES:
Ventilatory efficiency | Baseline (week 0), post-intervention (after 8 week intervention)
  Assessed via a maximal cardiopulmonary exercise test, using expired gas analysis under continuous electrocardiographic monitoring.
Heart rate dynamics | Baseline (week 0), post-intervention (after 8 week intervention)
  Assessed via 24-hour heart rate monitoring
Positive affect | Baseline (week 0), post-intervention (after 8 week intervention), 3 months post-intervention
  Positive and Negative Affect Schedule, a validated self-report measure, used to assess levels of positive affect. The positive affect subscale is made up of 10 items rated on a 5-point Likert scale. Scores range from 10 to 50 with higher scores indicating greater levels of positive affect
Emotion regulation | Baseline (week 0), post-intervention (after 8 week intervention), 3 months post-intervention
  Difficulties in Emotion Regulation Scale, a 36-item validated self-report measure, used to assess difficulties with emotion regulation; items are rated on a 5-point Likert scale, total scores range from 36 to 180, with higher scores reflecting greater emotion regulation difficulties. 6 subscale scores with higher scores reflecting greater emotion regulation difficulties.
Interoceptive awareness | Baseline (week 0), post-intervention (after 8 week intervention), 3 months post-intervention
  Multidimensional Assessment of Interoceptive Awareness Scale, a 32-item validated self-report measures, used to assess levels of interoceptive awareness; items are rated on a 6-point Likert scale, total scores range from 0 to 160, with higher scores reflecting greater interoceptive awareness. 8 subscales with higher scores reflecting greater interocpetive awareness
Self-efficacy | Baseline (week 0), post-intervention (after 8 week intervention), 3 months post-intervention
  Multidimensional Self-Efficacy Scale, a 9-item validated self-report measure, used to assess levels of self-efficacy; scores range from 0-90 with higher scores reflecting greater self-efficacy
Self-reported physical activity | Baseline (week 0), post-intervention (after 8 week intervention), 3 months post-intervention
  International Physical Activity Questionnaire, a validated self-report measure, used to assess levels of physical activity; walking MET mins/week, moderate MET mins/week and vigorous MET mins/week are calculated
Objective physical activity | Baseline (week 0), post-intervention (after 8 week intervention)
  7 day activity monitoring (via ActiGraph monitor) to assess minutes per week in moderate-intensity exercise
In-session oxygen consumption | Weeks 1 and 8
  Submaximal cardiopulmonary exercise testing (via standard metabolic cart)
In-session ventilatory efficiency | Weeks 1 and 8
  Submaximal cardiopulmonary exercise testing (via standard metabolic cart)
In-session respiration rate | Weeks 1 and 8
  Submaximal cardiopulmonary exercise testing (via standard metabolic cart)
In-session heart rate | Weeks 1 and 8
  Submaximal cardiopulmonary exercise testing (via standard metabolic cart)

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No